CLINICAL TRIAL: NCT02377661
Title: Lowering Blood Pressure in Primary Care in Vienna
Acronym: Low BP Vienna
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wilhelminenspital Vienna (Other)
Collaborators: Association for the Promotion of Research in Atherosclerosis, Thrombosis and Vascular Biology (Other); Ludwig Boltzmann Foundation for Cardiovascular Research (Unknown)
Responsible Party: Principal Investigator, Thomas Weiss, MD, PhD, MD, Wilhelminenspital Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V1-19012014
Record Dates: First submitted 2015-02-16; First posted 2015-03-03 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Treatment of hypertension according to current guidelines
- Experimental Care (Experimental): Treatment of hypertension using a standardised and simplified titration regime with single pill combinations, comprising an angiotensin receptor blocker, calcium channel blocker and hydrochlorothiazide.
  Interventions: Drug: Olmesartan medoxomil, amlodipine, hydrochlorothiazide

INTERVENTIONS:
Drug: Olmesartan medoxomil, amlodipine, hydrochlorothiazide — Up-titration of antihypertensive therapy with single pill combinations (comprising an angiotensin receptor blocker, calcium channel blocker and hydrochlorothiazide) in 4-week intervals if the target blood pressure of < 140/90 mmHg is not reached at the respective follow-up
  Arms: Experimental Care

SUMMARY:
The aim of this prospective, randomised, open-label, multicentre clinical trial is to enhance blood pressure control in primary care by introducing a standardised and simplified titration regime with single pill combinations (SPC), comprising an angiotensin receptor blocker, calcium channel blocker and hydrochlorothiazide.

DETAILED DESCRIPTION:
Rationale Hypertension is the single largest contributor to mortality worldwide, accounting for 13% of deaths globally. Approximately 30% of the adult population suffer from hypertension and of those diagnosed and treated, only 30-50% have adequately controlled blood pressure. At present, the importance of hypertension as fundamental risk factors is inadequately addressed among many patients and physicians.

Design The aim of this prospective, randomised, open-label, multicentre clinical trial is to enhance blood pressure control in primary care by introducing a standardised and simplified titration regime with single pill combinations (SPC), comprising an angiotensin receptor blocker, calcium channel blocker and hydrochlorothiazide.

The trial will randomise 42 family doctors or resident specialists for internal medicine (enrolling 840 patients with treated or untreated hypertension) to either experimental care or standard care for hypertension, latter according to the 2013 European Society of Cardiology Guidelines for the Management of Arterial Hypertension.

Practitioners randomised to experimental care will up-titrate antihypertensive therapy with SPCs in 4-week intervals if the target blood pressure of < 140/90 mmHg is not reached at the respective follow-up (Figure 1).

Study Outcomes The primary efficacy endpoint will be the proportion of patients achieving the target office blood pressure after 6 months of follow-up. The main secondary endpoint will be the improvement of 24h ambulatory blood pressure (ABPM) profile, measured at inclusion and after 6 months of follow-up.

Safety assessments include the evaluation of treatment emergent adverse events, particularly hospitalisation, worsening of renal function, peripheral oedema and hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* office blood pressure ≥ 140/90 mmHg
* ACE inhibitor intolerance (experimental arm)

Exclusion Criteria:

* Malignant disease with life expectancy < 6 months
* Women of childbearing potential (ICH definition) or breastfeeding
* Contraindications or allergies against olmesartan, amlodipine or hydrochlorothiazide (experimental arm)
* Chronic kidney disease grade IV or V (eGFR < 30 ml/min)
* Recent myocardial infarction or stroke within the preceding 3 months
* Participation in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Achievement of the target office blood pressure (< 140/90 mmHg) | 6 months
  Proportion of patients achieving the target office blood pressure of 140/90 mmHg
Achievement of the target systolic office blood pressure (< 140 mmHg) | 6 months
  Proportion of patients achieving the target systolic office blood pressure of 140 mmHg
Achievement of the target diastolic office blood pressure (< 90 mmHg) | 6 months
  Proportion of patients achieving the target diastolic office blood pressure of 90 mmHg

SECONDARY OUTCOMES:
Achievement of the target average 24h systolic ambulatory blood pressure (< 130 mmHg) | 6 months
  Average 24h systolic ambulatory blood pressure reading below 130 mmHg
Achievement of the target average 24h diastolic ambulatory blood pressure (< 80 mmHg) | 6 months
  Average 24h diastolic ambulatory blood pressure reading below 80 mmHg
Achievement of the target average daytime systolic ambulatory blood pressure (< 135 mmHg) | 6 months
  Average daytime systolic ambulatory blood pressure reading below 135 mmHg
Achievement of the target average nighttime systolic ambulatory blood pressure (< 120 mmHg) | 6 months
  Average nighttime systolic ambulatory blood pressure reading below 120 mmHg
Achievement of the target average daytime diastolic ambulatory blood pressure (< 85 mmHg) | 6 months
  Average daytime diastolic ambulatory blood pressure reading below 85 mmHg
Achievement of the target average nighttime diastolic ambulatory blood pressure (< 70 mmHg) | 6 months
  Average nighttime diastolic ambulatory blood pressure reading below 70 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Weiss, MD, PhD, Principal Investigator — 3rd Medical Department, Cardiology and Intensive Care Medicine Wilhelminenhospital, 1160 Vienna, Austria
Locations (1):
- GP practices, Vienna, Austria

REFERENCES:
- [Derived] Rohla M, Tscharre M, Huber K, Weiss TW. Lowering blood pressure in primary care in Vienna (LOW-BP-VIENNA) : A cluster-randomized trial. Wien Klin Wochenschr. 2018 Dec;130(23-24):698-706. doi: 10.1007/s00508-018-1374-4. Epub 2018 Aug 15. PMID 30112584